CLINICAL TRIAL: NCT00327431
Title: Relationship of Genes and Life Events to Blood Pressure
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Other Study IDs: 1000009109
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2008-05-22 (Estimated); Status verified 2008-05

CONDITIONS: Hypertension; Psychosocial Factors
Keywords: Hypertension; Blood Pressure; Psychosocial Factors
MeSH Terms: conditions — Hypertension | interventions — DNA

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Genetic: Cheek swab samples for DNA

SUMMARY:
Research suggests that blood pressure is influenced by both genetic and environmental factors. The goal of this study is to find genes that play a role in blood pressure and understand how they interact with life events (such as job stress) to influence blood pressure. We hypothesize that the gene for endothelin-1 is associated with increased blood pressure. Further, we predict that this genetic relationship is moderated by psychosocial stress factors, specifically job strain and marital cohesion.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in a study of psychosocial stressors and blood pressure (Double Exposure Study) and agreement to participate in follow-up studies

Exclusion Criteria:

* Withdrawal of consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2006-11; Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Baker, MB, ChB, Study Chair — University of Toronto; Sheldon Tobe, MD, Study Chair — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Tobe SW, Kiss A, Szalai JP, Perkins N, Tsigoulis M, Baker B. Impact of job and marital strain on ambulatory blood pressure results from the double exposure study. Am J Hypertens. 2005 Aug;18(8):1046-51. doi: 10.1016/j.amjhyper.2005.03.734. PMID 16109318